CLINICAL TRIAL: NCT06688461
Title: Effects of High Intensity Interval Training on Skeletal Muscle Insulin Sensitivity in Type 2 Diabetes Patients
Brief Title: High Intensity Interval Training and Insulin Sensitivity in Type 2 Diabetes
Acronym: T2D-HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finis Terrae University (Other)
Responsible Party: Principal Investigator, Rodrigo Mancilla, Doctor, PhD, Finis Terrae University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-001
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Lifestyle-related Condition; Insulin Sensitivity/Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Mental Disorders; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 1 interventional group of type 2 diabetes participants will undergo the 12-weeks of the HIIT program.
  1 non-interventional group of, age- and BMI matched, normoglycemic individuals will be the reference comparison for the post-training condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2D-HIIT (Experimental): This arm will perform HIIT under supervision. This arm will be compared to an age and BMI matched, normoglycemic non-intervention group.
  Interventions: Other: Experimental group: Exercise training
- NORM (No Intervention): This group of age-, BMI matched, normoglycemic individuals will the reference comparison for the T2D-HIIT arm post-intervention

INTERVENTIONS:
Other: Experimental group: Exercise training — HIIT program, 3 times per week for 12 weeks
  Arms: T2D-HIIT

SUMMARY:
A recognized driver for cardiovascular complications of type 2 diabetes mellitus (T2DM) is impaired plasma glucose homeostasis as consequence of skeletal muscle insulin resistance. Insulin-mediated plasma glucose disposal in skeletal muscle comprises oxidative glucose disposal (cellular glucose uptake for oxidation) and non-oxidative glucose disposal (NOGD; cellular glucose uptake for storage as glycogen), both processes being impaired in T2DM patients. Excessive intrahepatic fat accumulation (particularly monounsaturated (MUFA) and saturated (SFA)) is commonly observed in T2DM patients and tightly associates with plasma glucose dysregulation. It has been hypothesized that skeletal muscle insulin resistance redistributes circulating glucose away from muscle which together with hyperinsulinemia promotes intrahepatic lipid accretion via de novo lipogenesis (DNL). As saturated lipids is the final product of DNL, improving skeletal muscle insulin sensitivity, next to enhance plasma glucose homeostasis, might lower intrahepatic lipid content particularly intrahepatic saturated lipids.

Regular exercise is a cornerstone in the treatment of T2DM and to improve skeletal muscle insulin sensitivity. Interestingly, a conventional exercise program (aerobic-type combined with strength-type exercise) restores insulin-stimulated oxidative glucose disposal in T2DM patients to levels observed in age-matched normoglycemic subjects. Non-oxidative glucose disposal (NOGD), however, does not improve upon such conventional exercise programs. In this regard, for full restoration of compromised glucose disposal, it is pivotal to come up with effective training methods to target NOGD. High intensity interval training (HIIT) has the potential to expands the glycogen synthesis capacity in athletes by repetitive cycles of glycogen depletion/repletion, hence holds promise to improve NOGD in T2DM patients. Of note, HIIT also lowers the intrahepatic fat content in pre-diabetes individuals. Nevertheless, whether HIIT reduces the intrahepatic fat content and modifies its composition in T2DM patients is unknown. In this regard, it is hypothesized that HIIT expands the NOGD capacity in skeletal muscle of overweight/obese type 2 diabetes patients. By doing so, it is postulated that HIIT improves skeletal muscle insulin sensitivity and therefore benefits the 24 hours glycaemic profile in T2DM patients. In line, it is hypothesized that the HIIT-mediated improvements on NOGD and skeletal muscle insulin sensitivity coexist with the reduction of intrahepatic lipid content -particularly reduced saturated lipids- via lowering DNL.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Aged ≥ 45 and ≤ 75 years
* BMI: 25-35 kg/m2
* Diagnosed as T2DM patients for at least 1 year and not longer than 5 years
* HbA1c ≥ 6.5% and ≤ 8.5%
* Fasting blood glucose <130 mg/dL
* Women are post-menopausal (>1 year cessation of menses),
* Being stable on medication use of metformin and/or sulfonylurea derivatives for the previous 3 months or more and other medication naïve.

Exclusion Criteria:

* Type 1 diabetes
* Patients with congestive heart failure and and/or severe renal and or liver insufficiency
* Contraindications for MRI/MRS examination
* Active diabetic foot
* Polyneuropathy or retinopathy
* Signs of active liver or kidney dysfunction
* BMI >35 kg/m2
* Exogeneous insulin therapy
* Use of antidiabetic medication other than metformin or sulfonylurea derivatives treatment within 3 months before screening
* Use of SGLT2 inhibitors
* Unstable body weight (variations >5kg in the last 3 months)
* Ongoing weight loss diet or use of weight loss agents
* Uncontrolled hypertension
* Engagement in regular exercise program or any other medical condition that will impede the safe performance of the experiments

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin-stimulated non-oxidative plasma glucose disposal (NOGD) | 12 weeks
  Insulin-stimulated NOGD will be measured upon hyperinsulinemic-euglycemic clamp test

SECONDARY OUTCOMES:
Skeletal muscle insulin sensitivity | 12 weeks
  Skeletal muscle insulin sensitivity will be measured as the rate of insulin-stimulated plasma glucose disposal (Rd) measured upon hyperinsulinemic-euglycemic clamp test

OTHER OUTCOMES:
Insulin-stimulated glucose oxidation | 12 weeks
  Insulin-stimulated glucose oxidation will be measured via indirect calorimetry during clamp test
Metabolic flexibility | 12 weeks
  Metabolic flexibility will be measured via indirect calorimetry during the clamp test
Liver insulin sensitivity | 12 weeks
  Liver insulin sensitivity will be measured as the rate of insulin-mediated suppression of endogenous glucose production (EGP) upon hyperinsulinemic-euglycemic clamp test
24 hours glycemic profile | 12 weeks
  24 hours glycemic profile will be measured by the use of continuous glucose monitoring device
Intrahepatic lipid content and composition | 12 weeks
  Intrahepatic lipid content and composition will be measured by magnetic resonance spectroscopy of protons (1H-MRS)
De novo lipogenesis (DNL) | 12 weeks
  DNL will be measured by the use of deuterated water (D2O)
Skeletal muscle glycogen content | 12 weeks
  Muscle glycogen content will be quantified in muscle biopsies
Proteins that regulate oxidative metabolism | 12 weeks
  Content of proteins that regulate oxidative phosphorylation system (OXPHOS) will be quantified in muscle biopsies
Maximal aerobic capacity | 12 weeks
  Maximal aerobic capacity will be measure upon a progressive cycling test
Body weight | 12 weeks
  Body weight will be measured in kilograms
Total muscle mass | 12 weeks
  total muscle mass will be measured in kilograms and/or percentage
Total fat mass | 12 weeks
  Total fat mass will be measured in kilograms and/or percentage
Fat-free mass | 12 weeks
  Fat-free mass will be measured in kilograms and/or percentage
Skeletal muscle mutiomics | 12 weeks
  multiomics will be applied in muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Mancilla, PhD, Principal Investigator — Finis Terrae University
Locations (1):
- Finis Terrae University, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No